CLINICAL TRIAL: NCT03075904
Title: A Phase 1B/2, Multicenter, Open-Label, Safety, and Dose-Finding Study of SYNT001 in Subjects With Pemphigus (Vulgaris or Foliaceus)
Brief Title: A Safety and Dose-Finding Study of SYNT001 in Subjects With Pemphigus (Vulgaris or Foliaceus)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study objectives achieved
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYNT001-103
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Pemphigus; Pemphigus Vulgaris; Pemphigus Foliaceus
MeSH Terms: conditions — Pemphigus | interventions — orilanolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: ALXN1830 (Experimental): Participants received 5 doses of ALXN1830 10 mg/kg administered weekly.
  Interventions: Drug: ALXN1830
- Cohort 2: ALXN1830 (Experimental): Participants were to receive 3 doses of ALXN1830 30 mg/kg administered weekly (loading) followed by 5 doses of ALXN1830 10 mg/kg administered every other week or 10 weekly doses of ALXN1830 IV (maintenance).
  Interventions: Drug: ALXN1830

INTERVENTIONS:
Drug: ALXN1830 — Administered via IV infusion.
  Other Names: SYNT001

SUMMARY:
This was a multicenter, open-label safety study to determine the dose regimen of SYNT001 (ALXN1830) administered intravenously in participants with pemphigus (vulgaris or foliaceus).

DETAILED DESCRIPTION:
This study planned to evaluate 2 cohorts: up to 8 participants to receive 5 weekly intravenous (IV) doses of ALXN1830 at 10 milligram/kilogram (mg/kg) (Cohort 1) and up to 12 participants to receive 3 x 30 mg/kg weekly doses of ALXN1830 IV (loading) followed by 5 x 10 mg/kg doses of ALXN1830 IV every other week or 10 weekly doses of ALXN1830 IV (maintenance) (Cohort 2).

This study was terminated after the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy were characterized in participants with pemphigus at a single dose level (10 mg/kg) in Cohort 1, before any participants were enrolled in Cohort 2.

The study consisted of 3 periods: Screening, Treatment, and Follow-Up.

ELIGIBILITY:
Inclusion Criteria:

Participants must have meet the following criteria to be included:

* Were willing and able to read, understand and sign an informed consent form
* Documented diagnosis of pemphigus vulgaris or foliaceus
* Were required to use medically acceptable contraception

Exclusion Criteria:

Participants meeting any of the following criteria were excluded:

* Were unable or unwilling to comply with the protocol
* Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ)
* Positive for human immunodeficiency virus (HIV) or hepatitis C antibody
* Positive for hepatitis B surface antigen
* IV immunoglobulin treatment within 30 days of screening
* Any exposure to an investigational drug or device within the 30 days prior to screening
* Plasmapheresis or immunoadsorption within 30 days of screening
* Participant had any current medical condition that, in the opinion of the Investigator, may have compromised their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Alexion Study Site, Chapel Hill, North Carolina
  - Alexion Study Site, Durham, North Carolina
  - Alexion Study Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Werth VP, Culton DA, Concha JSS, Graydon JS, Blumberg LJ, Okawa J, Pyzik M, Blumberg RS, Hall RP 3rd. Safety, Tolerability, and Activity of ALXN1830 Targeting the Neonatal Fc Receptor in Chronic Pemphigus. J Invest Dermatol. 2021 Dec;141(12):2858-2865.e4. doi: 10.1016/j.jid.2021.04.031. Epub 2021 Jun 12. PMID 34126109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated after the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy were characterized at a single dose level (10 milligram/kilogram [mg/kg]) in Cohort 1, before any participants were enrolled in Cohort 2. This results disclosure is for Cohort 1 only.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1830
Started | 8
Received at Least 1 Dose of Study Drug | 8
Completed (All 8 participants received all 5 weekly doses of ALXN1830 10 mg/kg in the Treatment Period.) | 4
Not Completed | 4
Not completed — Physician Decision | 3
Not completed — Need for Medication not Permitted | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (16.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Type of Pemphigus [Count of Participants; unit: Participants]
  Vulgaris | 7
  Foliaceus | 1
Age at Diagnosis of Pemphigus [Mean (Standard Deviation); unit: years] | 41.3 (18.90)

OUTCOME MEASURES:

1. Primary Outcome: Count Of Participants Reporting Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) that starts on or after the first dose of study drug or occurs prior to the first dose and worsens in severity on or after the first dose of study drug, during the Treatment Period and Follow-up Period. A TEAE was considered "serious" (Grade 3) if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: death, life-threatening adverse drug event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, or an event that may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the previously listed outcomes. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1 (after first dose) through Day 112
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
Participants
  TEAEs | 7
  Serious TEAEs | 1
  Discontinuations due to TEAEs | 0
  Deaths | 0

2. Secondary Outcome: Maximum Percent Reduction Of Mean Total Immunoglobulin G (IgG) Levels From Baseline
Description: Pharmacodynamic samples were collected for analysis throughout the study. The maximum percent reduction of mean serum total IgG levels from Baseline observed during the study is presented.
Time Frame: Baseline through Day 112
Population: All participants who received at least 1 dose of study drug and had postdose pharmacodynamic data available.
Measure: Number; unit: percentage of reduction
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
percentage of reduction | 57.3

3. Secondary Outcome: Maximum Percent Reduction In Mean Pemphigus Disease Area Index (PDAI) Total Activity Score From Baseline
Description: Pemphigus severity and disease activity was measured using the PDAI in regions where a validated questionnaire was available. The PDAI was administered during Treatment Period and Follow-up Period. PDAI total activity was comprised of scores for the skin, mucous membrane, and scalp subscales. The investigator determined a PDAI score as 0 to 250 points for total activity score (0 to 120 for skin, 0 to 10 for scalp, and 0 to 120 for mucosa). A higher score indicated higher impact on skin disease. The maximum percent reduction in PDAI total activity score from Baseline observed during the study is presented.
Time Frame: Baseline through Day 112
Population: All participants who received at least 1 dose of study drug and had postdose pharmacodynamic data available.
Measure: Number; unit: percentage of reduction
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
percentage of reduction | 45.7

4. Secondary Outcome: Maximum Percent Reduction Of Mean Circulating Immune Complexes (CIC) Levels From Baseline
Description: Pharmacodynamic samples were collected for analysis throughout the study. The maximum percent reduction of mean CIC levels from Baseline observed during the study is presented.
Time Frame: Baseline through Day 112
Population: All participants who received at least 1 dose of study drug and had postdose pharmacodynamic data available.
Measure: Number; unit: percentage of reduction
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
percentage of reduction | 51.4

5. Secondary Outcome: Maximum Percent Reduction Of Mean Anti-Desmoglein (Dsg) 1 And 3 Antibodies From Baseline
Description: Pharmacodynamic samples were collected for analysis throughout the study. The maximum percent reduction of mean anti-Dsg 1 and 3 antibodies from Baseline observed during the study is presented.
Time Frame: Baseline through Day 112
Population: All participants who received at least 1 dose of study drug and had postdose pharmacodynamic data available.
Measure: Number; unit: percentage of reduction
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
percentage of reduction
  anti-Dsg 1 | 8.9
  anti-Dsg 3 | 20.4

ADVERSE EVENTS:
Time Frame: Baseline through Day 112
Arm/Group | Cohort 1: ALXN1830
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ALXN1830 (N=8)
Disease progression (General disorders) | 1 — Resolved and was considered to be not related to the study drug by the Investigator.
Acute kidney injury (Renal and urinary disorders) | 1 — Resolved and was considered to be not related to the study drug by the Investigator.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ALXN1830 (N=8)
Dry eye (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 1
Herpes simplex (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Tinea barbae (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Urine analysis abnormal (Investigations) | 1
Headache (Nervous system disorders) | 6
Sinus headache (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pallor (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is less than or equal to 60 days from the date that the communication is submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03075904/SAP_000.pdf
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT03075904/Prot_001.pdf